205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan | |
|---|---|---|
| Detailed Title: | An observational, retrospective, database study of the burden of seasonal Influenza A and B in Panama, selected countries of Central America and the Caribbean from the Year 2010 to 2015. | |
| eTrack study number and<br>Abbreviated Title | 205049 (EPI- | FLU-052 BOD PA DB) |
| Scope: | All data perta | ining to the above study. |
| Date of Statistical Analysis<br>Plan | 20-Sep-2017 | |
| Co-ordinating author: | PPD (Statistician) | |
| Reviewed by: | (Regional Epidemiologist) | |
| | PPD | (Director Epidemiology) |
| | (Lead statistician) | |
| | (Lead statistical analyst) | |
| | (Scientific writer) | |
| | PPD (Public disclosure representative) | |
| | (stat peer reviewer) | |
| Approved by: | PPD | (Regional Epidemiologist) |
| | PPD | (Lead statistician) |
| | PPD | (Scientific writer) |
| | PPD | (Lead statistical analyst) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIA | TIONS | 9 |
| 1. | DOCU | IMENT HI | STORY | 10 |
| 2. | STUD | Y DESIGI | N | 10 |
| 3. | OBJE0<br>3.1.<br>3.2. | Primary | objectiveary objectives | 11 |
| 4. | ENDP<br>4.1.<br>4.2. | Primary | endpointary endpoints | 11 |
| 5. | ANAL`<br>5.1. | Definition 5.1.1. 5.1.2. | S | 12<br>12 |
| 6. | STATI<br>6.1. | | ANALYSESaphyAnalysis of demographics/baseline characteristics planned in the protocol | 12 |
| | 6.2. | 6.1.2.<br>Primary<br>6.2.1.<br>6.2.2. | Additional considerations | 12<br>13<br>13 |
| | 6.3. | | Analysis of secondary objectives planned in the protocol Additional considerations | 13 |
| 7. | ANAL` | YSIS INTE | ERPRETATION | 13 |
| 8. | COND<br>8.1.<br>8.2. | Sequenc | ANALYSESe of analysesal considerations for interim analyses | 14 |
| 9. | CHAN | GES FRO | DM PLANNED ANALYSES | 14 |
| 10. | LIST | OF FINAL | REPORT TABLES, LISTINGS AND FIGURES | 15 |
| 11. | METH<br>11.1. | ODS<br>Statistica | IDARD DATA DERIVATION RULE AND STATISTICAL | 16 |
| | 11.2. | 11.2.1.<br>11.2.2. | d data derivation GSK legacy Date derivation Demography Case definition | 16 |

| | | 205049 (EPI-FLU-052 BOD PA DB) |
|---|---|---|
| | | Statistical Analysis Plan Final |
| 11.2.4. | Number of decimals displayed: | 17 |
| 12. ANNEX 2: SUM | IMARY ON ELIMINATION CODES | 17 |

## 205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## **LIST OF TABLES**

| | | PAGE |
|---------|---------------------------------------------|------|
| Table 1 | Study group and epoch foreseen in the study | 10 |

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Distribution of influenza positive specimens among number of specimen samples tested by calendar year - <country> (Screened cohort)</country> | 18 |
| Figure 2 | Distribution of influenza types among number of specimen samples tested by calendar year - <country> (Screened cohort)</country> | 19 |
| Figure 3 | Distribution of influenza positive specimens among number of specimen samples tested by influenza season - <country> (Screened cohort)</country> | 19 |
| Figure 4 | Distribution of influenza types among number of specimen samples tested by influenza season - <country> (Screened cohort)</country> | 19 |
| Figure 5 | Distribution of influenza types by age group - <country> (Total cohort)</country> | 24 |
| Figure 6 | Distribution of influenza A sub types by age group - <country> (Total cohort)</country> | 25 |
| Figure 7 | Distribution of influenza B lineage by age group - <country> (Total cohort)</country> | 26 |
| Figure 8 | Distribution of influenza types by region - <country> (Total cohort)</country> | 27 |
| Figure 9 | Distribution of influenza A subtypes by region - <country> (Total cohort)</country> | 28 |
| Figure 10 | Distribution of influenza B lineage by region - <country> (Total cohort)</country> | 29 |
| Figure 11 | Distribution of Influenza caused by influenza A and/or B among all influenza cases by calendar year - <country> (Total cohort)</country> | 31 |
| Figure 12 | Distribution of Influenza caused by influenza A and/or B among all influenza cases by influenza season - <country> (Total cohort)</country> | 31 |
| Figure 13 | Distribution of Influenza A subtypes among all influenza cases by calendar year - <country> (Total cohort)</country> | |
| Figure 14 | Distribution of Influenza A subtypes among all influenza cases by influenza season - <country> (Total cohort)</country> | |
| Figure 15 | Distribution of Influenza B lineage among all influenza cases by calendar year - <country> (Total cohort)</country> | 34 |

| | Statistical Analysis Plan Fina |
|---|---|
| Figure 16 | Distribution of Influenza B lineage among all influenza cases by influenza season - <country> (Total cohort)34</country> |
| Figure 17 | Circulation of influenza B lineage by season and recommended vaccine composition - <country> (Total cohort)38</country> |

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Number of specimen samples by calendar year - <country> (Screened cohort)</country> | 18 |
| Template 2 | Number of specimen samples by influenza season - <country> (Screened cohort)</country> | 19 |
| Template 3 | Summary of demographic characteristics by influenza types - <country> (Total cohort)</country> | 20 |
| Template 4 | Summary of demographic characteristics by influenza A subtypes and B lineages - <country> (Total cohort)</country> | 21 |
| Template 5 | Distribution of influenza A cases by month and year - <country> (Total cohort)</country> | 22 |
| Template 6 | Distribution of influenza B cases by month and year - <country> (Total cohort)</country> | 22 |
| Template 7 | Distribution of influenza A subtype H1N1 cases by month and year - <country> (Total cohort)</country> | 22 |
| Template 8 | Distribution of influenza A subtype H3N2 cases month and year - <country> (Total cohort)</country> | 23 |
| Template 9 | Distribution of influenza B lineage Victoria cases by month and year - <country> (Total cohort)</country> | 23 |
| Template 10 | Distribution of influenza B lineage Yamagata cases by month and year - <country> (Total cohort)</country> | 23 |
| Template 11 | Summary of influenza types by age group - <country> (Total cohort)</country> | 24 |
| Template 12 | Summary of influenza A subtypes by age group - <country> (Total cohort)</country> | 25 |
| Template 13 | Summary of influenza B lineage by age group - <country> (Total cohort)</country> | 26 |
| Template 14 | Summary of influenza types by region - <country> (Total cohort)</country> | 27 |
| Template 15 | Summary of influenza A subtypes by region - <country> (Total cohort)</country> | 28 |
| Template 16 | Summary of influenza B lineage by region - <country> (Total cohort)</country> | 29 |
| Template 17 | Proportion of Influenza caused by influenza A and/or B among all influenza cases by calendar year - <country> (Total cohort)</country> | 30 |

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

| Template 18 | Proportion of Influenza caused by influenza A and/or B among all influenza cases by influenza season - <country> (Total cohort)</country> | 30 |
|---|---|---|
| Template 19 | Proportion of Influenza A subtypes among all influenza cases by calendar year - <country> (Total cohort)</country> | 31 |
| Template 20 | Proportion of Influenza A subtypes among all influenza cases by influenza season - <country> (Total cohort)</country> | 32 |
| Template 21 | Proportion of Influenza B lineage among all influenza cases by calendar year - <country> (Total cohort)</country> | 33 |
| Template 22 | Proportion of Influenza B lineage among all influenza cases by influenza season - <country> (Total cohort)</country> | . 33 |
| Template 23 | Comparison of influenza B virus vaccine lineage and circulating lineage in the population by influenza season - <country> (Total cohort)</country> | 34 |
| Template 24 | Summary of signs and symptoms by influenza types and influenza season - <country> (Total cohort)</country> | 35 |
| Template 25 | Summary of signs and symptoms by influenza A subtypes and B lineage and influenza season - <country> (Total cohort)</country> | 37 |
| Template 26 | Summary of co-morbidity conditions by influenza types and influenza season- <country> (Total cohort)</country> | 38 |
| Template 27 | Summary of co-morbidity conditions by influenza A subtypes and B lineage and influenza season- <country> (Total cohort)</country> | 40 |
| Template 28 | Summary of treatments by influenza types and influenza season-<br><country> (Total cohort)</country> | 41 |
| Template 29 | Summary of treatments by influenza A subtypes and B lineage and influenza season - <country> (Total cohort)</country> | 41 |
| Template 30 | Summary of outcome by influenza types and influenza season-<br><country> (Total cohort)</country> | 42 |
| Template 31 | Summary of outcome by influenza A subtypes and B lineage - <country> (Total cohort)</country> | 42 |
| Template 32 | Summary of background information by influenza types - <country> (Total cohort)</country> | 43 |
| Template 33 | Summary of background information by influenza A subtypes and B lineage - <country> (Total cohort)</country> | 43 |

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

#### **LIST OF ABBREVIATIONS**

CI Confidence Interval

CTRS Clinical Trial Registry Summary

DB Database

GSK GlaxoSmithKline

ICGES Instituto Conmemorativo Gorgas de Estudios de la Salud

LL Lower Limit of the confidence interval

N.A. Not Applicable

SAP Statistical Analysis Plan

SD Standard Deviation

SLIPE Sociedad Latinoamericana de Infectología Pediátrica

SR Study Report

TFL Tables Figures and Listings
TIV Trivalent Influenza Vaccines

TOC Table of Content

UL Upper Limit of the confidence interval

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|--------------------------------|
| 20-SEP-2017 | Final version | Final Version 1: 29 March 2016 |

#### 2. STUDY DESIGN

- Type of study: Self-contained.
- Type of design: Epidemiological, non-interventional, observational, retrospective, database study.
- Study population: All subjects who have laboratory confirmed diagnosis of influenza (laboratory confirmed case) and reported in the national influenza surveillance system in selected countries from the Year 2010-2015.
- General study aspects: All seasonal influenza A and/or B cases reported in the ICGES database will be screened. Demographic data, date of onset of the first symptom and data on A-virus subtype and B-strain lineage, geographic region where the virus was isolated, clinical features and outcomes (clinical symptoms, duration of illness, complications) experienced by all influenza positive subjects (subjects with a laboratory confirmed influenza diagnosis) will be validated, extracted and transferred from the ICGES database to the sponsor or to the site of analysis, as applicable.
- Period of data collection: The study will include data on all the subjects with a laboratory confirmed influenza diagnosis, reported in the ICGES database of Panama, from January 2010 to December 2015. For all eligible subjects, individual level anonymised and key coded data will be collected from the database.
  - Epoch 001: Retrospective data collection.

Table 1 Study group and epoch foreseen in the study

| Study Group | Epoch |
|---------------|-----------|
| Study Group | Epoch 001 |
| Retrospective | X |

#### 3. OBJECTIVES

## 3.1. Primary objective

• To describe seasonal influenza A and/or B cases by age and virus subtype (AH1N1/A H3N2) and B-strain lineage (Victoria and Yamagata) using data reported via National Surveillance Program in Panama, selected countries of Central America and the Caribbean from January 2010 to December 2015.

## 3.2. Secondary objectives

From January 2010 to December 2015, in each selected country:

- To describe clinical features and outcomes (clinical manifestations, duration of illness, complications) of seasonal Influenza A and B cases in (overall and by subtypes or lineages) different seasons.
- To describe the temporal and geographical distribution of seasonal influenza A and/or B (overall and by subtypes or lineages) cases within different seasons.
- To estimate the percentage of co-circulation of influenza B lineages (Yamagata and Victoria lineages) among the study population, by age categories and by region.
- To describe the mismatch between the B-strain included in the Trivalent Influenza Vaccines (TIV) and the circulating B strains in different seasons.

#### 4. ENDPOINTS

## 4.1. Primary endpoint

• Occurrence of seasonal influenza A and/or B cases by age, virus subtype and strain lineage from the January 2010 to December 2015, in Panama, selected countries of Central America and the Caribbean (using the data reported via National Influenza Surveillance Program).

## 4.2. Secondary endpoints

- Occurrence of clinical features and outcomes (clinical symptoms, duration of illness, complications) experienced by subjects who have laboratory confirmed diagnosis seasonal influenza A and/or B, in different seasons from 2010 to 2015.
- Frequency of seasonal influenza A and/or B cases reported in different temporal and geographical locations within different seasons from 2010 to 2015.
- Occurrence of influenza caused by B-strain and presented by B lineages among the study population, by age (<1, 1-4, 5-9, 10-14, 15-19, 20-24, 25-44, 45-49, 50-59, 60-64 and  $\geq$  65 years) and by region.
- Compare the characteristics of the influenza B-infection as observed in the database and the B-strain included in the trivalent influenza vaccine.

#### 5. ANALYSIS SETS

#### 5.1. Definition

#### 5.1.1. Screened cohort

The screened cohort will include all the specimen samples received per year within the ICGES influenza surveillance system for influenza testing at aggregated level

#### 5.1.2. Total cohort

The Total cohort will comprise of all eligible subjects included in the study.

## 5.2. Criteria for eliminating data from Analysis Sets

Not applicable for database studies

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in annex 1 and will not be repeated below.

All the analysis on primary and secondary objectives will be performed on Total cohort.

## 6.1. Demography

## 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age and gender) will be summarised by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as gender.
- Mean, median and standard deviation will be provided for continuous data such as age.
- The distribution of influenza cases by month and year will also be tabulated.

#### 6.1.2. Additional considerations

Number of specimen samples received per year within the ICGES influenza surveillance system for influenza testing will be tabulated using frequency and percentages by calendar year and by Southern Hemisphere/Northern Hemisphere influenza season

### 6.2. Primary objective

#### 6.2.1. Analysis of primary objective planned in the protocol

The proportion of subjects with influenza caused by seasonal influenza A and/or B among all influenza cases reported with exact 95% confidence interval (CI) by age, A-virus subtype and B-strain lineage and overall will be calculated.

#### 6.2.2. Additional considerations

None

### 6.3. Secondary objectives

#### 6.3.1. Analysis of secondary objectives planned in the protocol

Seasonal influenza A and/or B cases will be described using frequency and percentages by temporal (calendar weeks/months) and geographical distributions (by country and by region within the country [if data is available]) within different influenza seasons (2010-2011, 2011-2012, 2012-2013, 2013-2014 and 2014-2015). Frequency and percentage for clinical features and outcomes (clinical manifestations, duration of illness, complications) experienced by influenza positive subjects will be tabulated by type of influenza (seasonal influenza A and/or B) in different seasons from 2010-2015. Frequency and percentage for influenza B lineages by age (<1, 1-4, 5-9, 10-14, 15-19, 20-24, 25-44, 45-49, 50-59, 60-64 and ≥ 65 years) and region will also be provided.

The characteristics of the influenza B-infection as observed in the database and the B strain included in the trivalent influenza vaccine will be assessed using frequency and percentage for each year. The proportion of matched B-strains and mis-matched B-strains will be estimated along with 95% CI.

#### 6.3.2. Additional considerations

Influenza A and/or B specimens (overall and by subtypes or lineages) will be described using frequency and percentages by country as well as Southern Hemisphere or Northern Hemisphere influenza season (depending which hemisphere influenza season the country follows). Example: Panama, El Salvador, Trinidad are considered as southern hemisphere and Guatemala, Dominican republic as northern hemisphere.

The proportion of mismatched B lineage will be calculated as 1 minus proportion of matched B lineage and expressed as percentages.

#### 7. ANALYSIS INTERPRETATION

All the analyses with respect to the primary and secondary endpoints will be descriptive. These descriptive analyses will not be interpreted, except describing the study results.

#### 8. CONDUCT OF ANALYSES

### 8.1. Sequence of analyses

There will be an interim analysis perform on available data (lab database for Panama) to submit the abstract/poster to SLIPE congress with preliminary results. The final analysis will be performed when all required data for the study have been extracted from the ICGES database and transferred to the sponsor or to the site of analysis, as applicable.

| Description | Analysis<br>ID | Disclosure Purpose (CTRS=public posting, SR=study report, internal) | Dry run<br>review<br>needed<br>(Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Analysis for<br>abstract/poster<br>submission to<br>SLIPE<br>congress | E1_01 | Abstract/poster submission | N | No | TFL TOC-<br>Abstract/poster<br>submission<br>(column J) |
| Final Analysis of epoch 1 | E1_02 | SR, CTRS | N | Yes | TFL TOC - All<br>TFLs |

## 8.2. Statistical considerations for interim analyses

All the analyses with respect to the primary and secondary endpoints will be descriptive/exploratory. As the results of the interim analyses will not be used to alter the study conduct, no statistical adjustment for interim analyses is required.

#### 9. CHANGES FROM PLANNED ANALYSES

- There will be an interim analysis planned on available data (lab database for Panama) in order to submit the abstract\poster for SLIPE congress
- We will also be reporting the number of specimen samples received per year within the ICGES influenza surveillance system for influenza testing at aggregated level (considered as screened cohort) and determine the proportion that tested positive for Influenza to describe the reporting capabilities of the surveillance system at capturing influenza A and B cases.
- We will also be including seasonal 2016 data as it is presently available. Based on the dates of data transfer, the end time period may be expanded if data is available during data transfer
- All the statistical analysis will be performed on specimens instead of subjects because a subject can provide more than one influenza positive specimens.
- The age group used for the analysis are 0-4, 5-17, 18-49, 50-64 and >=65 years instead of <1, 1-4, 5-9, 10-14, 15-19, 20-24, 25-44, 45-49, 50-59, 60-64 and  $\geq$  65 years.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The mock tables referred under column named 'layout' can be found in dedicated folder for standard tables and in Annex 3 for study specific mock table/figure/listing. The latter table/figure/listing are identified by the prefix SS\_ in the TFL Toc.

The following group names will be used in the TFLs:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| P | Influenza A | Positive for Influenza A |
| P | Influenza B | Positive for Influenza B |
| | Or/ar | nd |
| P | H1N1 | Positive for Influenza A subtype H1N1 |
| P | H3N2 | Positive for Influenza A subtype H3N2 |
| | Or/ar | nd |
| P | Victoria | Positive for Influenza B lineage Victoria |
| P | Yamagata | Positive for Influenza B lineage Yamagata |
| | Or/ar | nd |
| P | 0-4 | 0-4 years of age |
| P | 5-17 | 5-17 years of age |
| P | 18-49 | 18-49 years of age |
| P | 50-64 | 50-64 years of age |
| P | >=65 | >=65 years of age |
| | Or/ar | nd |
| P<br>P | West | West: Boca del Toro, Chiriquí and Comarca<br>Nobe Bugle |
| P<br>P | Central | Central: Coclé, Herrera, Los Santos and<br>Veraguas |
| P<br>P | Panama | Panamá: Panamá Este, Panamá Oeste,<br>Panamá Metro and San Miguelito |
| P<br>P | Northeast | Northeast: Colón, Darien and Kuna Yala |

| Influenza season | | |
|---|---|---|
| Calendar year (Jan-<br>Dec) | Southern Hemisphere (May-<br>Oct) | Northern Hemisphere (Oct-<br>May) |
| Jan-Dec 2010 | May- Oct 2010 | Oct 2010-May 2011 |
| Jan-Dec 2011 | May- Oct 2011 | Oct 2011-May 2012 |
| Jan-Dec 2012 | May- Oct 2012 | Oct 2012-May 2013 |
| Jan-Dec 2013 | May- Oct 2013 | Oct 2013-May 2014 |
| Jan-Dec 2014 | May- Oct 2014 | Oct 2014-May 2015 |
| Jan-Dec 2015 | May- Oct 2015 | Oct 2015-May 2016 |
| Jan-Dec 2016 | May- Oct 2016 | Oct 2016-May 2017 |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

- The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].
- WHO recommendations on the composition of influenza virus vaccines by influenza season can be found under: http://www.who.int/influenza/vaccines/virus/recommendations/en/

### 11.2. Standard data derivation GSK legacy

#### 11.2.1. Date derivation

• SAS date derived from a character date: In case day is missing, 15 is used. In case day & month are missing, 30June is used.

### 11.2.2. Demography

- Age at date of onset of the first symptom, will be expressed in years in the study. This will be computed as the difference between the date of onset of the first symptom and the date of birth (only if the data is available).
- The percentages will be computed by using only available information. Only frequencies will be provided for unknown or missing or not applicable categories
- Any measurements omitted or non-evaluable for a particular subject or analysis
  will not be replaced. Therefore, subjects with omitted or non-evaluable
  measurements will be excluded from the analysis

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

#### 11.2.3. Case definition

• Influenza is defined as any positive laboratory test from one or more of the clinical specimens [Guidelines for the epidemiological surveillance of influenza, 2012].

## 11.2.4. Number of decimals displayed:

The following decimal description from the decision rules will be used

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median age | 1 |
| Demographic characteristics | SD (age) | 1 |
| All summaries | % of count, including LL & UL of CI | 1 |

## 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Not Applicable

### 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following drafted study specific mocks will be used for each country (Panama, El Salvador, Guatemala and Trinidad, Dominican Republic, etc.,)

The data display, title and footnote is for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

Some these templates were copied from EPI-FLU-032 BOD MX DB (201075) study. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment

Template 1 Number of specimen samples by calendar year - <country> (Screened cohort)

| | Total specimen samples received | | Respiratory virus positive | | enza virus<br>ositive | enza A<br>itive | Influenza B positive | |
|---|---|---|---|---|---|---|---|---|
| Year | N | n | % | n | % | % | n | % |
| Jan-Dec 2010 | | | | | | | | |
| Jan-Dec 2011 | | | | | | | | |
| Jan-Dec 2012 | | | | | | | | |
| Jan-Dec 2013 | | | | | | | | |
| Jan-Dec 2014 | | | | | | | | |
| Jan-Dec 2015 | | | | | | | | |
| Jan-Dec 2016 | | | | | | | | |
| Total | | | | | | | | |

N =total number of specimen samples received

Figure 1 Distribution of influenza positive specimens among number of specimen samples tested by calendar year - <country> (Screened cohort)



n = number of positive specimen in a given category

<sup>%=(</sup>n/N)\*100

Figure 2 Distribution of influenza types among number of specimen samples tested by calendar year - <country> (Screened cohort)



Template 2 Number of specimen samples by influenza season - <country> (Screened cohort)

| | Total specimen samples received | | ratory<br>ositive | | ienza<br>positive | enza A<br>sitive | Influenza B positive | |
|---|---|---|---|---|---|---|---|---|
| <southern hemisphere="" influenza="" northern="" season=""></southern> | N | n | % | n | % | % | n | % |
| May- Oct 2010 | | | | | | | | |
| May- Oct 2011 | | | | | | | | |
| May- Oct 2012 | | | | | | | | |
| May- Oct 2013 | | | | | | | | |
| May- Oct 2014 | | | | | | | | |
| May- Oct 2015 | | | | | | | | |
| May- Oct 2016 | | | | | | | | |
| Total | | | | | | | | |

N =total number of specimen samples received

n = number of positive specimens in a given category

%=(n/N)\*100

Figure 3 Distribution of influenza positive specimens among number of specimen samples tested by influenza season - <country> (Screened cohort)

Refer to Figure 1

Figure 4 Distribution of influenza types among number of specimen samples tested by influenza season - <country> (Screened cohort)

Refer to Figure 2

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## Template 3 Summary of demographic characteristics by influenza types - <country> (Total cohort)

| | Parameters or Categories | | a A positive<br>N=XX | Influer | nza B positive<br>N=XX | Influenza virus posit<br>N = XX | |
|---|---|---|---|---|---|---|---|
| Characteristics | | Value or n | % | Value or n | % | Value or n | % |
| Age [Years] | n | | - | | - | | - |
| | Mean | | - | | - | | - |
| | SD | | - | | - | | - |
| | Median | | - | | - | | - |
| | Minimum | | - | | - | | - |
| | Maximum | | - | | - | | - |
| | Missing | | - | | - | | - |
| Age group [Years] | 0-4 | | | | | | |
| age group [Tears] | 5-17 | | | | | | |
| | 18-49 | | | | | | |
| | 50-64 | | | | | | |
| | >=65 | | | | | | |
| | Missing | | - | | - | | - |
| Gender | Female | | | | | | |
| | Male | | | | | | |
| Region | West | | | | | | |
| | Central | | | | | | |
| | Panama | | | | | | |
| | Northeast | | | | | | |
| Patient type | Outpatient | | | | | | |
| | Hospitalized | | | | | | |

N = number of influenza positive specimens

n = number of specimen positive in a given category

% = n / Number of specimens with available results x 100

Value = value of the considered parameter

SD = Standard deviation

West: Boca del Toro, Chiriquí and Comarca Nobe Bugle Central: Coclé, Herrera, Los Santos and Veraguas

Panamá: Panamá Este, Panamá Oeste, Panamá Metro and San Miguelito

Northeast: Colón, Darien and Kuna Yala

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## Template 4 Summary of demographic characteristics by influenza A subtypes and B lineages - <country> (Total cohort)

| | | | Influenza | A subtype | S | | Influenza B lineage | | |
|---|---|---|---|---|---|---|---|---|---|
| | Parameters or Categories | Н | 1N1<br>=XX | Н | 3N2<br>=XX | | ctoria<br>I=XX | Yamagat<br>N=XX | |
| Characteristics | | Value or n | % | Value or n | % | Value or n | % | Value or n | % |
| Age [Years] | n | | - | | - | | | | - |
| | Mean | | - | | - | | | | - |
| | SD | | - | | - | | | | - |
| | Median | | - | | - | | | | - |
| | Minimum | | - | | - | | | | - |
| | Maximum | | - | | - | | | | - |
| | Missing | | - | | - | | | | - |
| Age group [Years] | 0-4 | | | | | | | | |
| | 5-17 | | | | | | | | |
| | 18-49 | | | | | | | | |
| | 50-64 | | | | | | | | |
| | >=65 | | | | | | | | |
| | Missing | | - | | - | | | | - |
| Gender | Female | | | | | | | | |
| | Male | | | | | | | | |
| Region | West | | | | | | | | |
| · · | Central | | | | | | | | |
| | Panama | | | | | | | | |
| | Northeast | | | | | | | | |
| Patient type | Outpatient | | | | | | | | |
| •• | Hospitalized | | | | | | | | |

N = number of influenza positive specimens

n = number of specimen positive in a given category

% = n / Number of specimens with available results x 100

Value = value of the considered parameter

SD = Standard deviation

West: Boca del Toro, Chiriquí and Comarca Nobe Bugle Central: Coclé, Herrera, Los Santos and Veraguas

Panamá: Panamá Este, Panamá Oeste, Panamá Metro and San Miguelito

Northeast: Colón, Darien and Kuna Yala

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

Template 5 Distribution of influenza A cases by month and year - <country>
(Total cohort)

| Month and year<br>(date of onset of symptoms) | Influenza<br>virus positive<br>(N) | Influenza A<br>positive<br>(n) | Percentage (%) |
|---|---|---|---|
| Jan2010 | | • | |
| Feb2010 | | | |
| Mar 2010 | | | |
| Apr2010 | | | |
| May2010 | | | |
| Jun2010 | | | |
| Jul2010 | | | |
| Aug2010 | | | |
| Sep2010 | | | |
| Oct2010 | | | |
| Nov2010 | | | |
| Dec2010 | | | |
| Jan2011 | | | |
| Feb2011 | | | |
| Dec2016 | | | |

N = number of influenza positive specimens with available test results by month and year n = number of influenza A positive specimen in a given category  $% = (n / N) \times 100$ 

## Template 6 Distribution of influenza B cases by month and year - <country> (Total cohort)

Refer to Template 5

Template 7 Distribution of influenza A subtype H1N1 cases by month and year - <country> (Total cohort)

| Month and year<br>(date of onset of symptoms) | Influenza<br>virus positive<br>(N) | Influenza A<br>subtype H1N1<br>(n) | Percentage (%) |
|---|---|---|---|
| Jan2010 | , , | | |
| Feb2010 | | | |
| Mar 2010 | | | |
| Apr2010 | | | |
| May2010 | | | |
| Jun2010 | | | |
| Jul2010 | | | |
| Aug2010 | | | |
| Sep2010 | | | |
| Oct2010 | | | |
| Nov2010 | | | |
| Dec2010 | | | |
| Jan2011 | | | |
| Feb2011 | | | |
| Dec2016 | | | |

N = number of influenza positive specimens with available test results by month and year n = number of influenza A subtype H1N1 specimens in a given category % =  $(n / N) \times 100$ 

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## Template 8 Distribution of influenza A subtype H3N2 cases month and year - <country> (Total cohort)

Refer to Template 7

Template 9 Distribution of influenza B lineage Victoria cases by month and year - <country> (Total cohort)

| Month and year (date of onset of symptoms) | Influenza<br>virus positive<br>(N) | Influenza B<br>lineage Victoria<br>(n) | Percentage (%) |
|---|---|---|---|
| Jan2010 | | | |
| Feb2010 | | | |
| Mar 2010 | | | |
| Apr2010 | | | |
| May2010 | | | |
| Jun2010 | | | |
| Jul2010 | | | |
| Aug2010 | | | |
| Sep2010 | | | |
| Oct2010 | | | |
| Nov2010 | | | |
| Dec2010 | | | |
| Jan2011 | | | |
| Feb2011 | | | |
| Dec2016 | | | |

N = number of influenza positive specimens with available test results by month and year n = number of Influenza B lineage Victoria specimens in a given category % =  $(n / N) \times 100$ 

Template 10 Distribution of influenza B lineage Yamagata cases by month and year - <country> (Total cohort)

Refer to Template 9

Template 11 Summary of influenza types by age group - <country> (Total cohort)

| | | | 0-4<br>N=XX | | | | 5-17<br>N=XX | | | | <br>N=XX | | | | Total<br>N=XX | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Influenza type | Categories | n | % | % 95% | | n | n % | 95%<br>LL | 6 CI<br>UL | n | % | 95% CI<br>LL UL | | n | % | 95° | % CI |
| Influenza A | Positive | | | | UL | | | | - | | | | _ | | | | <u> </u> |
| | Negative | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - |
| Influenza B | Positive | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - |
| Influenza A and B | Both Positive | | | | | | | | | | | | | | | | |
| | Both Negative | | | | | | | | | | | | | | | | |
| | At least one positive | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - |

N = number of influenza positive specimens by age group

Figure 5 Distribution of influenza types by age group - <country> (Total cohort)



n = number of specimens in a given category

<sup>% =</sup> n / Number of specimens with available results x 100

<sup>95%</sup>CI= exact confidence interval; LL=lower limit; UL=upper limit

Template 12 Summary of influenza A subtypes by age group - <country> (Total cohort)

| | 0-4<br>N=XX | | | | | 5-17<br>N=XX | | | | N=XX | | | | Total<br>N=XX | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Influenza A sub- | Categories | n | % | 95% | CI | n | % | 95% | CI | n | % | 95% | CI | n | % | 95% | 6 CI |
| type | | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL |
| H1N1 | Positive | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - |
| H3N2 | Positive | | | | | | | | | | | | | | | | |
| <u> </u> | Negative | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - |

N = number of influenza positive specimens by age group

n = number of specimens in a given category

% = n / Number of specimens with available results x 100

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

Figure 6 Distribution of influenza A sub types by age group - <country> (Total cohort)



Template 13 Summary of influenza B lineage by age group - <country> (Total cohort)

| | | | 0-4<br>N=XX | | | | 5-17<br>N=XX | | | | N=XX | | | | Total<br>N=XX | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Influenza B lineage | Categories | n | % | 95% | CI | n | % | 95% CI | | n | % | 95% CI | | n | % | 95% | 6 CI |
| | | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL |
| Victoria | Positive | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - |
| Yamagata | Positive | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - |

N = number of influenza positive specimens by age group

n = number of specimens in a given category

% = n / Number of specimens with available results x 100

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

Figure 7 Distribution of influenza B lineage by age group - <country> (Total cohort)



Template 14 Summary of influenza types by region - <country> (Total cohort)

| | | | - | Vest<br>I=X) | | | | entra<br>I=X) | | | | nan<br>I=X) | | | | orth<br>N=) | east<br>(X | | Tota<br>N=X | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Influenza | Categories | n | % | 95% | % CI | n | % | 95% | 6 CI | n | % | 95 | % CI | n | % | 9 | 5% CI | n | % | 95% | % CI |
| type | | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL |
| Influenza A | Positive | | | | | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - | | - | - | - |
| Influenza B | Positive | | | | | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - | | - | - | - |
| Influenza A<br>and B | Both Positive | | | | | | | | | | | | | | | | | | | | |
| | Both Negative | | | | | | | | | | | | | | | | | | | | |
| | At least one positive | | | | | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - | | - | - | - |

N = number of influenza positive specimens by region

n = number of specimens in a given category

% = n / Number of specimens with available results x 100

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

West: Boca del Toro, Chiriquí and Comarca Nobe Bugle

Central: Coclé, Herrera, Los Santos and Veraguas

Panamá: Panamá Este, Panamá Oeste, Panamá Metro and San Miguelito

Northeast: Colón, Darien and Kuna Yala

Figure 8 Distribution of influenza types by region - <country> (Total cohort)



Template 15 Summary of influenza A subtypes by region - <country> (Total cohort)

| | | | | Vest | | | | ntra<br>=XX | | Pa | anar | na N | =XX | | | orthe<br>N=X | east<br>X | | Tota<br>N=X | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Influenza A | Categories | n | % | 95% | 6 CI | N | % | 95% | 6 CI | n | % | 959 | % CI | n | % | 95 | % CI | n | % | 95% | δ CI |
| subtypes | | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL |
| H1N1 | Positive | | | | | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - | | - | - | - |
| H3N2 | Positive | | | | | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | - | - | - | | - | - | - |

N = number of influenza positive specimens by age group

n = number of specimens in a given category

% = n / Number of specimens with available results x 100

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

West: Boca del Toro, Chiriquí and Comarca Nobe Bugle Central: Coclé, Herrera, Los Santos and Veraguas

Panamá: Panamá Este, Panamá Oeste, Panamá Metro and San Miguelito

Northeast: Colón, Darien and Kuna Yala

Figure 9 Distribution of influenza A subtypes by region - <country> (Total cohort)



Template 16 Summary of influenza B lineage by region - <country> (Total cohort)

| | | | | Ves<br>I=X) | | | | ntr<br>=X) | | Pa | naı | na N | =XX | | N | orth<br>N=X | | | Tota<br>N=XX | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Influenza B<br>lineage | Categories | n | % | | 5%<br>CI | N | % | | 5%<br>CI | n | % | 959 | % CI | n | % | 9 | 5% CI | n | % | | 5%<br>CI |
| | | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL | | | LL | UL |
| Victoria | Positive | | | | | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | | | | | - | - | - |
| Yamagata | Positive | | | | | | | | | | | | | | | | | | | | |
| | Negative | | | | | | | | | | | | | | | | | | | | |
| | Missing/Unknown | | - | - | - | | - | - | - | | - | - | - | | | | | | - | - | - |

N = number of influenza positive specimens by age group

n = number of specimens in a given category

% = n / Number of specimens with available results x 100

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

West: Boca del Toro, Chiriquí and Comarca Nobe Bugle

Central: Coclé, Herrera, Los Santos and Veraguas

Panamá: Panamá Este, Panamá Oeste, Panamá Metro and San Miguelito

Northeast: Colón. Darien and Kuna Yala

Figure 10 Distribution of influenza B lineage by region - <country> (Total cohort)



205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

Template 17 Proportion of Influenza caused by influenza A and/or B among all influenza cases by calendar year - <country> (Total cohort)

| | | | | | | 95% CI |
|---------------|----------------|---|---|---|----|--------|
| Calendar year | Influenza type | n | N | % | LL | UL |
| 2010 | Influenza A | | | | | |
| | Influenza B | | | | | |
| 2011 | Influenza A | | | | | |
| | Influenza B | | | | | |
| 2012 | Influenza A | | | | | |
| | Influenza B | | | | | |
| 2013 | Influenza A | | | | | |
| | Influenza B | | | | | |
| 2014 | Influenza A | | | | | |
| | Influenza B | | | | | |
| 2015 | Influenza A | | | | | |
| | Influenza B | | | | | |
| 2016 | Influenza A | | | | | |
| | Influenza B | | | | | |
| Total | Influenza A | | | | | |
| | Influenza B | | | | | |

N = Number of Influenza positive specimens with available test results by year

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

Template 18 Proportion of Influenza caused by influenza A and/or B among all influenza cases by influenza season - <country> (Total cohort)

| | | | | | 9 | 5% CI |
|---|---|---|---|---|---|---|
| <southern hemisphere<br="" northern="">Influenza season&gt;</southern> | Influenza type | n | N | % | LL | UL |
| May- Oct 2010 | Influenza A | | | | | |
| · | Influenza B | | | | | |
| May- Oct 2011 | Influenza A | | | | | |
| • | Influenza B | | | | | |
| May- Oct 2012 | Influenza A | | | | | |
| • | Influenza B | | | | | |
| May- Oct 2013 | Influenza A | | | | | |
| · | Influenza B | | | | | |
| May- Oct 2014 | Influenza A | | | | | |
| • | Influenza B | | | | | |
| May- Oct 2015 | Influenza A | | | | | |
| • | Influenza B | | | | | |
| May- Oct 2016 | Influenza A | | | | | |
| • | Influenza B | | | | | |
| Total | Influenza A | | | | | |
| | Influenza B | | | | | |

N = Number of Influenza positive specimens with available test results by year

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

n = Number of positive specimens in a given category

<sup>% = (</sup>n/N) \* 100

n = Number of positive specimens in a given category

 $<sup>% = (</sup>n/N)^* 100$ 

Figure 11 Distribution of Influenza caused by influenza A and/or B among all influenza cases by calendar year - <country> (Total cohort)



Figure 12 Distribution of Influenza caused by influenza A and/or B among all influenza cases by influenza season - <country> (Total cohort)

Refer to Figure 11

Template 19 Proportion of Influenza A subtypes among all influenza cases by calendar year - <country> (Total cohort)

| | | | | | | 95% CI |
|-------|----------------------|---|---|---|----|--------|
| Year | Influenza A subtypes | n | N | % | LL | UL |
| 2010 | H1N1 | | | | | |
| | H3N2 | | | | | |
| 2011 | H1N1 | | | | | |
| | H3N2 | | | | | |
| 2012 | H1N1 | | | | | |
| | H3N2 | | | | | |
| 2013 | H1N1 | | | | | |
| | H3N2 | | | | | |
| 2014 | H1N1 | | | | | |
| | H3N2 | | | | | |
| 2015 | H1N1 | | | | | |
| | H3N2 | | | | | |
| 2016 | H1N1 | | | | | |
| | H3N2 | | | | | |
| Total | H1N1 | | | | | |
| | H3N2 | | | | | |

N = Number of Influenza positive specimens with available test results by year

n = Number of positive specimens in a given category

% = n/N \* 100

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

Template 20 Proportion of Influenza A subtypes among all influenza cases by influenza season - <country> (Total cohort)

| | | | | | | 95% CI |
|---|---|---|---|---|---|---|
| <southern northern<br="">hemisphere influenza season&gt;</southern> | Influenza A subtypes | n | N | % | LL | UL |
| May- Oct 2010 | H1N1 | | | | | |
| | H3N2 | | | | | |
| May– Oct 2011 | H1N1 | | | | | |
| | H3N2 | | | | | |
| May- Oct 2012 | H1N1 | | | | | |
| | H3N2 | | | | | |
| May- Oct 2013 | H1N1 | | | | | |
| | H3N2 | | | | | |
| May- Oct 2014 | H1N1 | | | | | |
| | H3N2 | | | | | |
| May- Oct 2015 | H1N1 | | | | | |
| · | H3N2 | | | | | |
| May- Oct 2016 | H1N1 | | | | | |
| - | H3N2 | | | | | |
| Total | H1N1 | | | | | |
| | H3N2 | | | | | |

N = Number of Influenza positive specimens with available test results by year

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

Figure 13 Distribution of Influenza A subtypes among all influenza cases by calendar year - <country> (Total cohort)



Figure 14 Distribution of Influenza A subtypes among all influenza cases by influenza season - <country> (Total cohort)

Refer to Figure 13

n = Number of positive specimens in a given category

<sup>% =</sup> n/N \* 100

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## Template 21 Proportion of Influenza B lineage among all influenza cases by calendar year - <country> (Total cohort)

| | | | | | | 95% CI |
|-------|---------------------|---|---|---|----|--------|
| Year | Influenza B lineage | n | N | % | LL | UL |
| 2010 | Victoria | | | | | |
| | Yamagata | | | | | |
| 2011 | Victoria | | | | | |
| | Yamagata | | | | | |
| 2012 | Victoria | | | | | |
| | Yamagata | | | | | |
| 2013 | Victoria | | | | | |
| | Yamagata | | | | | |
| 2014 | Victoria | | | | | |
| | Yamagata | | | | | |
| 2015 | Victoria | | | | | |
| | Yamagata | | | | | |
| 2016 | Victoria | | | | | |
| | Yamagata | | | | | |
| Total | Victoria | | | | | |
| | Yamagata | | | | | |

N = Number of Influenza positive specimens with available test results by year

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

Template 22 Proportion of Influenza B lineage among all influenza cases by influenza season - <country> (Total cohort)

| | | | | | | 95% CI |
|---|---|---|---|---|---|---|
| <southern hemisphere="" influenza="" northern="" season=""></southern> | Influenza B lineage | n | N | % | LL | UL |
| May- Oct 2010 | Victoria | | | | | |
| | Yamagata | | | | | |
| May- Oct 2011 | Victoria | | | | | |
| · | Yamagata | | | | | |
| May- Oct 2012 | Victoria | | | | | |
| · | Yamagata | | | | | |
| May- Oct 2013 | Victoria | | | | | |
| · | Yamagata | | | | | |
| May- Oct 2014 | Victoria | | | | | |
| · | Yamagata | | | | | |
| May- Oct 2015 | Victoria | | | | | |
| • | Yamagata | | | | | |
| May- Oct 2016 | Victoria | | | | | |
| - | Yamagata | | | | | |
| Total | Victoria | | | | | |
| | Yamagata | | | | | |

N = Number of Influenza positive specimens with available test results by year

95%CI= exact confidence interval; LL=lower limit; UL=upper limit

n = Number of positive specimens in a given category

<sup>% =</sup> n/N \* 100

n = Number of positive specimens in a given category

<sup>% =</sup> n/N \* 100

Figure 15 Distribution of Influenza B lineage among all influenza cases by calendar year - <country> (Total cohort)



Figure 16 Distribution of Influenza B lineage among all influenza cases by influenza season - <country> (Total cohort)

Refer to Figure 15

Template 23 Comparison of influenza B virus vaccine lineage and circulating lineage in the population by influenza season - <country> (Total cohort)

| <southern hemisphere="" influenza="" northern="" season=""></southern> | Circulating lines | Influen<br>ages | za B | Vaccine Recommendation* | %<br>Match | % |
|---|---|---|---|---|---|---|
| innuenza season> | B lineage | n | % | Recommendation | waten | Mismatch |
| 2010 | Victoria | | | Victoria | | |
| 2010 | Yamagata | | | Victoria | | |
| 2011 | Victoria | | | Victoria | | |
| 2011 | Yamagata | | | Victoria | | |
| 2012 | Victoria | | | Victoria | | |
| 2012 | Yamagata | | | Victoria | | |
| 2013 | | | | Yamagata | | |
| 2014 | | | | Yamagata | | |
| 2015 | | | | | | |
| 2016 | | | | | | |

<sup>\*</sup>http://www.who.int/influenza/vaccines/virus/recommendations/en/

n = Number of influenza positive specimens in a given category

<sup>% =</sup> n / Number of specimens with available results x 100

<sup>%</sup> Mismatch = 100% - % Circulating B lineage match with vaccine

Figure 17 Circulation of influenza B lineage by season and recommended vaccine composition - <country> (Total cohort)



Template 24 Summary of signs and symptoms by influenza types and influenza season - <country> (Total cohort)

| | | | A po | enza<br>sitive<br>XX | pos | nza B<br>itive<br>XX | po | luenza<br>virus<br>ositive<br>= XX |
|---|---|---|---|---|---|---|---|---|
| <pre><southern hemisphere="" influenza="" northern="" season=""></southern></pre> | Signs and symptoms | Categories | n | % | n | % | n | % |
| May- Oct 2010 | Sudden onset of | Yes | | | | | | |
| | symptoms | No | | | | | | |
| | | Unknown | | - | | - | | |
| | Fever | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Malice | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Cough | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Rhinorrhea | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | | | | | |
| | Headache | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Polypnea | Yes | | | | | | |
| | | No | | | | | | _ |
| | | Unknown | | - | | - | | - |

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

| | | | Influenza<br>A positive<br>N=XX | | Influenza<br>virus<br>positive<br>N = XX |
|---|---|---|---|---|---|
| | Dyspnea | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | - |
| | Vomiting | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | - |
| | Myalgia | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | - |
| | Arthralgia | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | - |
| | Irritability | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | - |
| | Odynophagia | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | - |
| | Abdominal pain | Yes | | | |
| | · | No | | | |
| | | Unknown | - | - | - |
| | Diarrhea | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | - |
| | Conjunctivitis | Yes | | | |
| | | No | | | |
| | | Unknown | - | - | |
| | Chest pain | Yes | | | |
| | Citost pain | No | + + | † † | |
| | | Unknown | | - | _ |
| | Cyanosis | Yes | + + | † † | |
| | 5,4,100,0 | No | + + | † † | |
| | | Unknown | | - | - |
| | Chills | Yes | <del> </del> | <del> </del> | |
| | Ottillo | No | <del> </del> | <del> </del> | |
| | | Unknown | <del> </del> | - | - |
| May- Oct 2011 | | CHRIOWII | | + + - | |
| May- Oct 2012 | | | + + | + + | |
| • | | | | | |
| | | | + + | + + | |
| <br>Total | | | | + | |

N = number of influenza positive specimens by groups n = number of positive specimens in a given category % = n / Number of subjects with available results x 100

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

# Template 25 Summary of signs and symptoms by influenza A subtypes and B lineage and influenza season - <country> (Total cohort)

| | | | ; | ıflue<br>subt | уре | S | | lin | enza<br>eage | ! |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Yam<br>N= | agata<br>-XX |
| <southern northern<br="">hemisphere influenza<br/>season&gt;</southern> | Signs and symptoms | Categories | n | % | n | % | n | % | n | % |
| May- Oct 2010 | Sudden onset of | Yes | | | | | | | | |
| | symptoms | No | | | | | | | | |
| | , | Unknown | | | | | | - | | - |
| | Fever | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Malice | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Cough | Yes | | | | | | | | |
| | Jougn | | | | | | | | | |
| | | No<br>Unknown | | | | | | _ | | _ |
| | Rhinorrhea | Yes | | | | | | | | |
| | Headache | No | | | | | | | | |
| | | Unknown | | | | | | | | |
| | | Yes | | | | | | | | |
| | riodddono | No | | | | | | | | |
| | | Unknown | | | | | | _ | | _ |
| | Polypnea | Yes | | | | | | | | |
| | i olypnod | No | | | | | | | | |
| | | Unknown | | | | | | _ | | _ |
| | Dyspnea | Yes | | | | | | | | |
| | Буорной | No | | | | | | | | |
| | | Unknown | | | | | | _ | | - |
| | Vomiting | Yes | | | | | | | | |
| | Volimang | No | | | | | | | | |
| | | Unknown | | | | | | _ | | _ |
| | Myalgia | Yes | | | | | | | | |
| | iviyaigia | No | | | | | | | | |
| | | Unknown | - | | | | | _ | | _ |
| | Arthralgia | Yes | | | | | | <del>-</del> | | - |
| | / www.aigia | No | | | | | | | | |
| | | Unknown | - | | | | | _ | | _ |
| | Irritability | Yes | | | | | | <del> -</del> | | <del>-</del> |
| | Irritability | No | | | | | | | | |
| | | | - | | | | | | | |
| | | Unknown | | | | | | - | | - |

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

| | | | | | | | | | | II FIIIa |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | lue | | | | Influ | | |
| | | | | | | S | | | eage | |
| | | | | | | | | | | agata |
| | | | N=X | XX | N= | XX | N=XX | | N= | =XX |
| | Odynophagia | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Abdominal pain | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Diarrhea | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Conjunctivitis | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Chest pain | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Cyanosis | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| | Chills | Yes | | | | | | | | |
| | | No | | | | | | | | |
| | | Unknown | | | | | | - | | - |
| May- Oct 2011 | | | | | | | | | | |
| May- Oct 2012 | | | | | | | | | | |
| Total | | | | | | | | | | |
| VI | scitive encoimens by groups | | | | | | | | | |

Template 26 Summary of co-morbidity conditions by influenza types and influenza season- <country> (Total cohort)

| | | | ро | enza A<br>sitive<br>=XX | Influenza B<br>positive<br>N=XX | | Influenza<br>virus positive<br>N = XX | |
|---|---|---|---|---|---|---|---|---|
| <southern hemisphere="" influenza="" northern="" season=""></southern> | Co-morbidity condition | Categories | n | % | n | % | n | % |
| May- Oct 2010 | Diabetes | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Chronic obstructive | Yes | | | | | | |
| | pulmonary disease | No | | | | | | |
| | (COPD) | Unknown | | - | | - | | - |
| | Asthma | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |

N = number of influenza positive specimens by groups n = number of positive specimens in a given category % = n / Number of specimens with available results x 100

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

| | | | | ıza A<br>tive | Influ<br>po | enza B<br>sitive<br>=XX | Infl<br>virus | uenza<br>positive<br>= XX |
|---|---|---|---|---|---|---|---|---|
| <southern hemisphere="" influenza="" northern="" season=""></southern> | Co-morbidity condition | Categories | n | % | n | % | n | % |
| | Inmunosuppression | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Hypertension | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | HIV/AIDS | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Cardiovascular disease | Yes | | | | 1 | | |
| | | No | | | | <del> </del> | | |
| | | Unknown | | _ | | - | | _ |
| | Obesity | Yes | | | | | | |
| | No<br>Unk | | | | | | | |
| | | Unknown | | _ | | 1_ | | _ |
| | | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Chronic renal failure | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Pregnancy | Yes | | | | | | |
| | 3 3 3 | No | | | | | | |
| | | Unknown | | - | | - | | - |
| | Months of pregnancy | n | | _ | | _ | | _ |
| | | Mean | | - | | - | | - |
| | | SD | | - | | - | | - |
| | | Median | | - | | - | | - |
| | | Minimum | | - | | - | | - |
| | | Maximum | | - | | - | | - |
| | | N.A./Unknown | | - | | - | | - |
| May- Oct 2011 | | | | | | | | |
| Total | | | | | | | | |

N = number of influenza positive specimens by groups
n = number of influenza positive specimens in a given category
% = n / Number of specimens with available results x 100

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

# Template 27 Summary of co-morbidity conditions by influenza A subtypes and B lineage and influenza season- <country> (Total cohort)

| | | | | Influe<br>sub | enza<br>type: | | Inf | luenz | a B lineage |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 1N1<br>=XX | НЗ | 3N2<br>=XX | | toria<br>=XX | Yamagata<br>N=XX |
| <southern northern<br="">hemisphere influenza season&gt;</southern> | Co-morbidity condition | Categories | n | % | n | % | n | % | |
| May- Oct 2010 | Diabetes | Yes | | | | | | | |
| • | | No | | | | | | | |
| | | Unknown | | - | | - | | - | |
| | Chronic obstructive | Yes | | | | | | | |
| | pulmonary disease | No | | | | | | | |
| | (COPD) | Unknown | | - | | - | | - | |
| | Asthma | Yes | | | | | | | |
| | | No | | | | | | | |
| | | Unknown | | - | | - | | - | |
| | Inmunosuppression | Yes | | | | | | | |
| | | No | | | | | | | |
| | | Unknown | | - | | - | | _ | |
| | Hypertension | Yes | | | | | | | |
| | 7,600.000 | No | | | | | | | |
| | | Unknown | | - | | - | | _ | |
| | HIV/AIDS | Yes | | | | | | | |
| | THV// NDC | No | | | | | | | |
| | | Unknown | | _ | | | | | |
| | Cardiovascular disease | Yes | | | | | | | |
| | Cardiovasculai disease | No | | | | | | | |
| | | Unknown | | | | | | | |
| | Obesity | Yes | | - | | | | - | |
| | Obesity | No | | | | | | | |
| | | Unknown | | | | | | | |
| | Smoking | 1 | | - | | - | | - | |
| | Smoking | Yes<br>No | | | | | | | |
| | | Unknown | | | | | | | |
| | Chronic renal failure | | | - | | - | | - | |
| | Chronic renai fallure | Yes | | | | | | | |
| | | No | | | | | | | |
| | D | Unknown | | - | | - | | - | |
| | Pregnancy | Yes | | | | | | | |
| | | No | | | | | | | |
| | | Unknown | | - | | - | | - | |
| | Months of pregnancy | n | | - | | - | 1 | - | |
| | | Mean | | - | | - | | - | |
| | | SD | | - | 1 | - | 1 | - | |
| | | Median | | - | | - | | - | |
| | | Minimum | | - | | - | | - | |
| | | Maximum | | - | | - | | - | |
| | | N.A./Unknown | | - | | - | | - | |
| May- Oct 2011 | | | | | | | | | |
| | | | | | $\perp$ | | $\perp$ | | |
| Total | | | | 1 | | | | | |

N = number of influenza positive specimens by groups

n = number of positive specimens in a given category % = n / Number of specimens with available results x 100

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

#### Template 28 Summary of treatments by influenza types and influenza season-<country> (Total cohort)

| | | | pos | Influenza A<br>positive<br>N=XX | | enza B<br>sitive<br>=XX | Influenza viru<br>positive<br>N = XX | |
|---|---|---|---|---|---|---|---|---|
| <southern hemisphere="" influenza="" northern="" season=""></southern> | Treatment | Categories | n | % | n | % | n | % |
| May- Oct 2010 | Treatment received | Yes | | | | | | |
| | from the beginning of | No | | | | | | |
| | <i>'</i> ' | Unknown | | - | | - | | - |
| | | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown/NA | | - | | - | | - |
| | Microbial Treatment | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown/NA | | - | | - | | - |
| May- Oct 2011 | | | | | | | | |
| Total | | | | | | | | |

N = number of influenza positive specimens by groups

Template 29 Summary of treatments by influenza A subtypes and B lineage and influenza season - <country> (Total cohort)

| | | | Influ | ıenza | A sub | types | Influenza | B lineage |
|---|---|---|---|---|---|---|---|---|
| | | | | N1<br>XX | | 3N2<br>=XX | Victoria<br>N=XX | Yamagata<br>N=XX |
| <southern northern<br="">hemisphere influenza season&gt;</southern> | Treatment | Categories | n | % | n | % | n | % |
| May- Oct 2010 | Treatment received | Yes | | | | | | |
| - | from the beginning | No | | | | | | |
| | of symptoms | Unknown | | - | | - | | |
| | | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown/NA | | - | | - | | |
| | Microbial Treatment | Yes | | | | | | |
| | | No | | | | | | |
| | | Unknown/NA | | - | | - | | |
| May- Oct 2011 | | | | | | | | |
| Total | | | | | | | | |

N = number of influenza positive specimens by groups

n = number of positive specimens in a given category

<sup>% =</sup> n / Number of specimens with available results x 100

n = number of positive specimens in a given category

<sup>% =</sup> n / Number of specimens with available results x 100

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

### Template 30 Summary of outcome by influenza types and influenza season-<country> (Total cohort)

| | | pos | enza A<br>sitive<br>=XX | pos | enza B<br>sitive<br>=XX | pos | za virus<br>sitive<br>= XX |
|---|---|---|---|---|---|---|---|
| <southern northern<br="">hemisphere influenza season&gt;</southern> | Outcome | n | % | n | % | n | % |
| May- Oct 2010 | Discharged | | | | | | |
| • | Serious case | | | | | | |
| | No serious case | | | | | | |
| | Death | | | | | | |
| | Missing | | - | | - | | - |
| May- Oct 2011 | | | | | | | |
| Total | | | | | | | |

N = number of influenza positive specimens by groups

Template 31 Summary of outcome by influenza A subtypes and B lineage - <country> (Total cohort)

| | | In | fluenza | A subty | pes | Inf | luenza l | B lineage | |
|---|---|---|---|---|---|---|---|---|---|
| | | | IN1<br>=XX | | N2<br>XX | Vict<br>N= | - | | agata<br>XX |
| <southern hemisphere="" influenza="" northern="" season=""></southern> | Outcome | n | % | n | % | n | % | n | % |
| May- Oct 2010 | Discharged | | | | | | | | |
| | Serious case | | | | | | | | |
| | No serious case | | | | | | | | |
| | Death | | | | | | | | |
| | Missing | | - | | - | | | | - |
| May- Oct 2011 | | | | | | | | | |
| Total | | | | | | | | | |

N = number of influenza positive specimens by groups

n = number of positive specimens in a given category

<sup>% =</sup> n / Number of specimens with available results x 100

n = number of positive specimens in a given category

<sup>% =</sup> n / Number of specimens with available results  $\dot{x}$  100

205049 (EPI-FLU-052 BOD PA DB) Statistical Analysis Plan Final

## Template 32 Summary of background information by influenza types - <country> (Total cohort)

| | | pos | enza A<br>itive<br>XX | Influenza B<br>positive<br>N=XX | | pos | za virus<br>itive<br>: XX |
|---|---|---|---|---|---|---|---|
| History | Categories | n | % | n | % | n | % |
| Previous contact with other influenza | Yes | | | | | | |
| cases | No | | | | | | |
| | Missing | | - | | - | | - |
| Previous contact with Birds | Yes | | | | | | |
| | No | | | | | | |
| | Missing | | - | | - | | - |
| Previous contact with Pigs | Yes | | | | | | |
| · · | No | | | | | | |
| | Missing | | - | | - | | - |
| Previous contact with other animals | Yes | | | | | | |
| | No | | | | | | |
| | Missing | | - | | - | | - |
| Previous vaccination against seasonal nfluenza | Yes | | | | | | |
| | No | | | | | | |
| | Missing | | - | | - | | - |

N = number of influenza positive specimens by groups

Template 33 Summary of background information by influenza A subtypes and B lineage - <country> (Total cohort)

| | | Infl | uenza A | subty | pes | Ir | ıfluenza | B lineag | ge |
|---|---|---|---|---|---|---|---|---|---|
| | | | 1N1<br>=XX | | 3N2<br>=XX | Victoria<br>N=XX | | Yama<br>N= | |
| History | Categories | n | % | n | % | n | % | n | % |
| Previous contact with other | Yes | | | | | | | | |
| influenza cases | No | | | | | | | | |
| | Missing | | - | | - | | | | |
| Previous contact with Birds | Yes | | | | | | | | |
| | No | | | | | | | | |
| | Missing | | - | | - | | | | |
| Previous contact with Pigs | Yes | | | | | | | | |
| | No | | | | | | | | |
| | Missing | | - | | - | | | | |
| Previous contact with other | Yes | | | | | | | | |
| animals | No | | | | | | | | |
| | Missing | | - | | - | | | | |
| Previous vaccination against | Yes | | | | | | | | |
| seasonal influenza | No | | | | | | | | |
| | Missing | | - | | - | | | | |

N = number of influenza positive specimens by groups

n = number of positive specimens in a given category

<sup>% =</sup> n / Number of specimens with available results x 100

n = number of positive specimens in a given category

<sup>% =</sup> n / Number of specimens with available results x 100